CLINICAL TRIAL: NCT03090048
Title: Treatment of Acne for Cases Resistant to Currently Available Measures Via Vitamin A With or Without Azithromycin in Topical Formulations
Brief Title: Vitamin A and Azithromycin for Acne Vulgaris
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manchanda Medical Clinic (Other)
Responsible Party: Principal Investigator, DR. VINOD C TAWAR, Principal investigator, Manchanda Medical Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tawar -1
Record Dates: First submitted 2017-01-29; First posted 2017-03-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Vitamin A; retinol palmitate; Azithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin A (Experimental): retinyl palmitate USP
  Interventions: Drug: Vitamin A
- Azithromycin with Vitamin A (Experimental): USP grade ingredients
  Interventions: Drug: Vitamin A; Drug: Azithromycin
- Azithromycin (Active Comparator): azithromycin monohydrate
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Vitamin A — Vitamin A 2-3 % concentration
  Other Names: retinyl palmitate
  Arms: Azithromycin with Vitamin A; Vitamin A
Drug: Azithromycin — azithromycin monohydrate
  Other Names: azithromycin monohydrate
  Arms: Azithromycin; Azithromycin with Vitamin A

SUMMARY:
Patients seen with acne lesions not having responded to existing treatments will be offered a placebo or a topical preparation consisting of Vitamin A USP with or without Azithromycin for a duration of 4-6 months USP for the objective of resolving the lesions without systemic side effects and via weekly follow-ups.

DETAILED DESCRIPTION:
The concentrations of the active ingredients is based on the enclosed articles and the formulations have been modified with an objective of minimizing the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active lesions

Exclusion Criteria:

* Patients on a treatment
* Asymptomatic patients

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-08-24 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Measurement (dimensions) of acne lesions | Every 4 weeks up to16 weeks
  follow-up focussed on observation of changes

CONTACTS AND LOCATIONS:
Overall Officials: Vinod C Tawar, Study Director — M.D.
Locations (1):
- Manchanda Mc, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bartlett KB, Davis SA, Feldman SR. Tolerability of topical antimicrobials in treatment of acne vulgaris. J Drugs Dermatol. 2014 Jun;13(6):658-62. PMID 24918554